CLINICAL TRIAL: NCT01331798
Title: Clinical Evaluation of the Cohera TissuGlu Device in the Management of Wound Drainage Following Abdominoplasty
Brief Title: Evaluation of Cohera TissuGlu in the Management of Wound Drainage Following Abdominoplasty
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Contact: Chad Coberly, VP Clinical Affairs, Cohera Medical Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-100-0002
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Abdominoplasty
Keywords: Abdominoplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test: TissuGlu Adhesive (Experimental): Patients received the TissuGlu Adhesive Treatment
  Interventions: Device: Cohera TissuGlu Surgical Adhesive
- Control (Active Comparator): Control Arm received no TissuGlu- Standard of Care received.
  Interventions: Procedure: Control- Standard of care

INTERVENTIONS:
Device: Cohera TissuGlu Surgical Adhesive — TissuGlu device used prior to closing of the flap in the abdominoplasty procedure.
  Arms: Test: TissuGlu Adhesive
Procedure: Control- Standard of care — Control Arm- no TissuGlu device used. Standard abdominoplasty procedure followed.
  Arms: Control

SUMMARY:
A blinded, prospective, randomized trial in 40 abdominoplasty cases at three sites to study the safety and the preliminary efficacy of TissuGlu®, a novel surgical adhesive, in the management of wound drainage during abdominoplasty procedures.

DETAILED DESCRIPTION:
Background: Fluid accumulation in dissected tissue planes has been a longstanding problem following surgical procedures. The common use of closed suction drains has been associated with infection risk, wound healing complications, additional scarring, and patient discomfort. Additionally, seroma formation after drain removal often requires invasive treatment. Therapies that can reduce fluid accumulation and decrease the need for drains will have a positive impact on surgical practice.

Objective: To study the safety and the preliminary efficacy of a TissuGlu®, a novel surgical adhesive, in the management of wound drainage during abdominoplasty procedures.

Material & Methods: A blinded prospective randomized trial compared drain fluid output (volume) and complication profile in 40 subjects undergoing abdominoplasty with (n=20) or without (n=20) the use of a urethane based adhesive. The TissuGlu® adhesive, which required no mixing or preparation, was administered to the abdominal wall using a custom drop tip applicator prior to closure of the abdominoplasty flap. Two Blake® drains connected to J-VAC suction reservoirs were placed in the wound.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 20 years of age;
* Be in good general health in the opinion of the Investigator with no conditions that would significantly impact wound healing as determined by medical history and review of recent concomitant medications;
* Be scheduled for at least one full thickness surgical incision of at least 20cm in length as part of elective abdominoplasty requiring the placement of sutures in the superficial fascia and subcutaneous tissue to relieve skin tension prior to final skin closure, Surgeon must use electrocautery in the procedure;
* Be willing to follow instructions for incision care, comply with schedule for wound drainage volume measurements, and follow guidelines related to resumption of daily activities;
* Agree to return for all follow-up evaluations specified in this protocol;
* Agree not to schedule any additional elective surgical procedures that involve an incision until their participation in this study is complete; and
* Sign the informed consent.

Exclusion Criteria:

* Anesthesia Risk judged to be higher than ASA2
* Previous Abdominoplasty
* Have severe co-morbid conditions that pose a high risk for surgery and adequate recovery (e.g., heart disease)
* Any condition involving compromised vascular flow to the abdominal wall tissue. Prior abdominal scars, especially subcostal scars, will be a relative contraindication and judged on a case by case basis by the surgeon investigator.
* Any condition known to effect wound healing, such as collagen vascular disease
* Current active tobacco use, including smokeless (chewing) tobacco
* Obesity, as defined by BMI >30
* Known blood clotting disorder
* Current diagnosis of diabetes
* Be receiving antibiotic therapy for pre-existing condition or infection
* Have known personal or family history of keloid formation or hypertrophy
* Undergoing concurrent adjacent or congruent Liposuction procedures
* Concurrent use of fibrin sealants or other internal wound care devices
* Be currently taking systemic steroids or immunosuppressive agents
* Concurrent hernia repair greater than 6 cm and/or requiring the use of mesh
* Mini abdominoplasty (Abdominoplasty without umbilical transposition)
* Have known or suspected allergy or sensitivity to any test materials or reagents
* Be participating in any current clinical trial or have participated in any clinical trial within 30 days of enrollment in this study
* Pregnancy (30 days post-op)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
• Safety data will be gathered with respect to the number, timing, severity, duration and resolution of device and non-device related adverse events occurring among study subjects. | Discharge, 14, 30, 60, 90 Day follow-up

SECONDARY OUTCOMES:
• Time to drain removal based upon a drain removal criteria of <30ml of fluid accumulation in a twenty four (24) hour period (Scevola et al, 2002; Momeni et al, 2008). | Assessed at time of drain removal- Average 2 to 5 days post surgery.
• Number of wound complications, seroma formation, wound dehiscence, infection, skin necrosis, hematoma | Discharge, 14, 30, 60, 90 Day follow-up
• Cumulative drainage volume for each patient | Assessed at time of drain removal- Average 2-5 days post surgery.
• Number of additional physician or clinic visits | Discharge, 14, 30, 60, 90 Day follow-up
• Number/type of additional procedures due to complications | Discharge, 14, 30, 60, 90 Day follow-up
• Evaluation of the delivery method/delivery device (Surgeon questionnaire) | Assessed at time of surgery/use of the device (Day 0)
  Questionnaire completed by the surgeon after the surgery rating ergonomics, visibility, ability to deliver the adhesive and overall satisfaction with the delivery method.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University of Bonn, Bonn
  - Rosenpark Klinik, Darmstadt
  - Erich-Lexer-Klinik, Freiburg im Breisgau